CLINICAL TRIAL: NCT01829568
Title: A Phase I Study of Rituximab, Lenalidomide, and Ibrutinib in Previously Untreated Follicular Lymphoma
Brief Title: Rituximab, Lenalidomide, and Ibrutinib in Treating Patients With Previously Untreated Stage II-IV Follicular Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00792; NCI-2013-00792 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CALGB-A051103; A051103 (Other: Alliance for Clinical Trials in Oncology); A051103 (Other: CTEP); U10CA031946 (NIH); U10CA180821 (NIH)
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Ann Arbor Stage II Grade 1 Contiguous Follicular Lymphoma; Ann Arbor Stage II Grade 1 Non-Contiguous Follicular Lymphoma; Ann Arbor Stage II Grade 2 Contiguous Follicular Lymphoma; Ann Arbor Stage II Grade 2 Non-Contiguous Follicular Lymphoma; Ann Arbor Stage II Grade 3 Contiguous Follicular Lymphoma; Ann Arbor Stage II Grade 3 Non-Contiguous Follicular Lymphoma; Ann Arbor Stage III Grade 1 Follicular Lymphoma; Ann Arbor Stage III Grade 2 Follicular Lymphoma; Ann Arbor Stage III Grade 3 Follicular Lymphoma; Ann Arbor Stage IV Grade 1 Follicular Lymphoma; Ann Arbor Stage IV Grade 2 Follicular Lymphoma; Ann Arbor Stage IV Grade 3 Follicular Lymphoma
MeSH Terms: interventions — ibrutinib; Lenalidomide; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (lenalidomide, ibrutinib, and rituximab) (Experimental): Patients receive lenalidomide PO QD on days 1-21 and ibrutinib PO QD on days 1-28. Treatment repeats every 28 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV on days 1, 8, 15, and 22 of cycle 1 and once weekly at weeks 13, 21, 29, and 37.
  Interventions: Drug: Ibrutinib; Drug: Lenalidomide; Biological: Rituximab

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA 032765; CRA-032765; CRA032765; Imbruvica; PCI 32765; PCI-32765; PCI32765
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima

SUMMARY:
This phase I trial studies the side effects and best dose of lenalidomide and ibrutinib when given together with rituximab in treating patients with previously untreated stage II-IV follicular lymphoma. Lenalidomide may stimulate the immune system in different ways and stop cancer cells from growing. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Rituximab is a monoclonal antibody. It binds to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. Giving lenalidomide and ibrutinib together with rituximab may work well in treating follicular lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the recommended phase II doses of ibrutinib and lenalidomide for combination with rituximab in previously untreated follicular lymphoma.

SECONDARY OBJECTIVES:

I. To determine pharmacokinetics of ibrutinib and its major metabolite (PCI-45227) when combined with lenalidomide and rituximab.

II. To determine the pharmacodynamics of basophil activation and Bruton tyrosine kinase (BTK) occupancy in peripheral blood mononuclear cells (PBMCs) over a 24-hour period of ibrutinib when given in combination with lenalidomide and rituximab.

OUTLINE: This is a dose-escalation study of lenalidomide and ibrutinib.

Patients receive lenalidomide orally (PO) once daily (QD) on days 1-21 and ibrutinib PO QD on days 1-28. Treatment repeats every 28 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab intravenously (IV) on days 1, 8, 15, and 22 of cycle 1 and once weekly at weeks 13, 21, 29, and 37.

After completion of study treatment, patients are followed up every 4 months for 2 years and then every 6 months for 8 years or every 6 months or annually for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, histologically confirmed follicular lymphoma, World Health Organization (WHO) classification grade I, II, or IIIa (> 15 centroblasts per high power field with centrocytes present) that is stage III, IV, or bulky (i.e., single mass >= 7 cm in any unidimensional measurement) stage II and requires therapy at the discretion of the primary physician

  * Bone marrow biopsies as the sole means of diagnosis are not acceptable, but they may be submitted in conjunction with nodal biopsies; fine needle aspirates are not acceptable for diagnosis
  * Failure to submit pathology specimens within 60 days of patient registration will be considered a major protocol violation
  * Institutional flow cytometry or immunohistochemistry must confirm cluster of differentiation 20 (CD20) antigen expression
  * All risk by follicular lymphoma international prognostic index (FLIPI): 0-5 risk factors
* No prior systemic therapy for non-Hodgkin lymphoma (NHL) including chemotherapy or immunotherapy (e.g., monoclonal antibody-based therapy), radiation therapy, or radioimmunotherapy
* For non-NHL conditions, no chemotherapy, radiotherapy, or major surgery within 4 weeks (6 weeks for nitrosoureas or mitomycin C) of enrollment; no patients who have ongoing adverse events from agents administered more than 4 weeks previously
* No prior exposure to any of the study agents
* No corticosteroids within two weeks prior to study entry, except for maintenance therapy for a non-malignant disease; dose of corticosteroid or prednisone (or its equivalent) should not exceed 20 mg per day; corticosteroid premedication for rituximab is allowed
* Eastern Cooperative Oncology Group (ECOG) performance status must be =< 2
* Measurable disease must be present either on physical examination or imaging studies; non-measurable disease alone is not acceptable; any tumor mass > 1 cm is acceptable; lesions that are considered non-measurable include the following:

  * Bone lesions (lesions if present should be noted)
  * Ascites
  * Pleural/pericardial effusion
  * Lymphangitis cutis/pulmonis
  * Bone marrow (involvement by NHL should be noted)
* Patients with human immunodeficiency virus (HIV) infection are eligible, provided they meet the following:

  * No evidence of coinfection with hepatitis B or C
  * CD4+ cell count >= 400/mm^3
  * No evidence of resistant strains of HIV
  * If not on anti-HIV therapy, HIV viral load < 10,000 copies HIV ribonucleic acid (RNA)/mL
  * If on anti-HIV therapy, HIV viral load < 50 copies HIV RNA/mL
  * No history of acquired immunodeficiency syndrome (AIDS)-defining conditions
  * No use of strong cytochrome P450, family 3, subfamily A, polypeptide 4/5 (CYP3A4/5) inhibitors or inducers
* No known central nervous system (CNS) involvement by lymphoma
* No treatment with strong inhibitors or inducers of CYP3A4/5
* No evidence of active hepatitis B or C infections (i.e., no positive serology for anti-hepatitis B virus [HBV] or anti-hepatitis C virus [HCV] antibodies); HBV seropositive patients (hepatitis B surface antigen [HBsAg] +) are eligible if they are closely monitored for evidence of active HBV infection by HBV deoxyribonucleic acid (DNA) testing and receive suppressive therapy with lamivudine or other HBV suppressive therapy until 6 months after the last rituximab dose
* No history of erythema multiforme, toxic epidermal necrolysis or Stevens-Johnson syndrome
* No history of uncontrolled seizures
* No autoimmune disorder that requires active immunosuppression
* No intracranial hemorrhage within the last 6 months
* Patients must be non-pregnant and non-nursing; females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days and again within 24 hours prior to starting cycle 1 of lenalidomide; further, they must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy; a FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy, or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time preceding 24 consecutive months); all patients must be counseled by a trained counselor every 28 days about pregnancy precautions and risks of fetal exposure
* No known human anti-chimeric antibody (HACA) positivity
* No anticoagulation with warfarin is allowed; patients must not have received warfarin within 28 days prior to registration; alternative anticoagulant may be used
* Patients must not be receiving concurrent treatment with other investigational drugs
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to lenalidomide, ibrutinib, or other agents used in study
* Patients must not have presence of transfusion-dependent thrombocytopenia
* No currently active clinically significant cardiovascular disease including the following:

  * No uncontrolled arrhythmia
  * No congestive heart failure
  * No class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
  * No history of myocardial infarction, deep venous or arterial thrombosis within 6 months prior to registration
* No prior malignancy with the exceptions listed below:

  * Malignancy treated with curative intent and with no evidence of active disease for more than 3 years prior to screening and felt to be at low risk for recurrence by the treating physician
  * Adequately treated non-melanomatous skin cancer or lentigo maligna melanoma without current evidence of disease
  * Adequately treated cervical carcinoma in situ without current evidence of disease
* Patients must be >= 18 years of age
* Absolute neutrophil count (ANC) >= 1,000/microliter (should be present independent of growth factor or transfusion support for at least 7 days prior to first dose of study drug)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN) (should be present independent of growth factor or transfusion support for at least 7 days prior to first dose of study drug)
* Total bilirubin =< 1.5 x ULN unless attributable to Gilbert's syndrome (should be present independent of growth factor or transfusion support for at least 7 days prior to first dose of study drug)
* Creatinine clearance > 60 mL/min (patients on dialysis are not eligible); to be calculated by method of Cockcroft-Gault, using actual weight (should be present independent of growth factor or transfusion support for at least 7 days prior to first dose of study drug)
* Creatinine =< 2 x ULN (should be present independent of growth factor or transfusion support for at least 7 days prior to first dose of study drug)
* Platelet count >= 75,000/microliter (should be present independent of growth factor or transfusion support for at least 7 days prior to first dose of study drug)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-06-26 (Actual); Primary Completion 2015-05-11 (Actual); Study Completion 2026-06-06 (Estimated)

PRIMARY OUTCOMES:
Maximally tolerated dose (MTD) of lenalidomide and ibrutinib for combination with rituximab | 28 days
  Defined as the highest dose at which 0 or 1 of 6 patients experience DLT. Will be determined by dose-limiting toxicities (DLT) graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

SECONDARY OUTCOMES:
Toxicities by attribute and grade | Up to 10 years
  Summarized for each dose level. Will be assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Complete response rate | Up to 10 years
  Estimated for each dose level.
Overall response rate | Up to 10 years
  Estimated for each dose level.
Progression-free survival (PFS) | The time between registration and disease progression or death, assessed up to 10 years
  Estimated by Kaplan-Meier method for the whole number of patients in this study and at the MTD.
Overall survival (OS) | The time between registration and death, assessed up to 10 years
  Estimated by Kaplan-Meier method for the whole number of patients in this study and at the MTD.

OTHER OUTCOMES:
Pharmacokinetic parameters of ibrutinib and major metabolite PCI-45227 | Days 1 and 15 of course 1 and week 13 (pre-dose, 1, 2, 4, 7, and 24 hours post-ibrutinib dose)
  Tabulated and summarized using descriptive statistics.
BTK parameters | At 4 hours and 24 hours post ibrutinib dosing
  Tabulated and summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Chaitra S Ujjani, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (7):
- United States (7):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- [Derived] Rutherford SC, Yin J, Pederson L, Perez Burbano G, LaPlant B, Shadman M, Li H, LeBlanc ML, Kenkre VP, Hong F, Blum KA, Dockter T, Martin P, Jung SH, Grant B, Rosenbaum C, Ujjani C, Barr PM, Unger JM, Cheson BD, Bartlett NL, Kahl B, Friedberg JW, Mandrekar SJ, Leonard JP. Relevance of Bone Marrow Biopsies for Response Assessment in US National Cancer Institute National Clinical Trials Network Follicular Lymphoma Clinical Trials. J Clin Oncol. 2023 Jan 10;41(2):336-342. doi: 10.1200/JCO.21.02301. Epub 2022 Jul 5. PMID 35787017
- [Derived] Ujjani CS, Jung SH, Pitcher B, Martin P, Park SI, Blum KA, Smith SM, Czuczman M, Davids MS, Levine E, Lewis LD, Smith SE, Bartlett NL, Leonard JP, Cheson BD. Phase 1 trial of rituximab, lenalidomide, and ibrutinib in previously untreated follicular lymphoma: Alliance A051103. Blood. 2016 Nov 24;128(21):2510-2516. doi: 10.1182/blood-2016-06-718106. Epub 2016 Oct 3. PMID 27697771